CLINICAL TRIAL: NCT01298882
Title: Effect of Diacerein on Insulin Secretion in Patients With Type 2 Diabetes Mellitus and Overweight or Obesity
Brief Title: Diacerein on Insulin Secretion in Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Collaborators: National Council of Science and Technology, Mexico (Other)
Responsible Party: Manuel González-Ortiz, CIS Mexico
Model: Parallel | Purpose: Treatment
Other Study IDs: DIADM2-001
Record Dates: First submitted 2011-01-31; First posted 2011-02-18 (Estimated); Last update posted 2011-02-18 (Estimated); Status verified 2011-01

CONDITIONS: Type 2 Diabetes Mellitus; Overweight; Obesity
Keywords: Type 2 diabetes mellitus; Overweight; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity | interventions — diacerein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diacerein (Experimental)
  Interventions: Drug: Diacerein
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Diacerein
  Arms: Diacerein
Other: Placebo
  Arms: Placebo

SUMMARY:
Aim. To assess the effect of interleukin 1β (IL-1β) and tumor necrosis factor α (TNFα) inhibition with diacerein administration on insulin secretion and metabolic control of drug-naïve patients with type 2 diabetes mellitus (T2DM) and overweight or obesity.

Hypothesis. Diacerein administration improves insulin secretion and metabolic control of drug-naïve patients with type 2 diabetes mellitus (T2DM) and overweight or obesity.

Materials and methods. Design: Randomized, double-blind, placebo-controlled clinical trial. Population: 40 drug-naïve adult patients with T2DM and overweight or obesity. Measurements: A metabolic profile including IL-1β, TNFα, interleukin 6, and fasting insulin levels, as well as, hyperglycemic-hyperinsulinemic clamp technique; to assess the phases of insulin secretion and insulin sensitivity. Intervention for 2 mo: diacerein (50 mg once daily) for the first 15 days and twice daily for 45 additional days or placebo. Statistical analyses: Wilcoxon signed rank and Mann-Whitney U test.

ELIGIBILITY:
Inclusion Criteria:

* Fasting glucose levels between 7.0 and 11.1 mmol/L
* A1C levels between 7 and 9%
* Same residential area and socioeconomic status
* Excessively sedentary or participated in heavy physical activity
* Nonsmokers
* Body weight was stable for at least 3 months before the study
* Blood pressure was <130/80 mm Hg

Exclusion Criteria:

* Personal history of hepatic, renal or coronary artery disease
* Medications known to affect metabolism during the previous 6 months.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult

PRIMARY OUTCOMES:
Fasting insulin concentration | 2 mo
Fasting glucose concentration | 2 mo
A1C concentration | 2 mo
First phase of insulin secretion | 2 mo
Late phase of insulin secretion | 2 mo
Total insulin secretion concentration | 2 mo

CONTACTS AND LOCATIONS:
Locations (1):
- Unidad de Investigación Médica en Epidemiología Clínica, Guadalajara, Jalisco, Mexico

REFERENCES:
- [Derived] Ramos-Zavala MG, Gonzalez-Ortiz M, Martinez-Abundis E, Robles-Cervantes JA, Gonzalez-Lopez R, Santiago-Hernandez NJ. Effect of diacerein on insulin secretion and metabolic control in drug-naive patients with type 2 diabetes: a randomized clinical trial. Diabetes Care. 2011 Jul;34(7):1591-4. doi: 10.2337/dc11-0357. Epub 2011 May 24. PMID 21610123